CLINICAL TRIAL: NCT04069741
Title: Treating Depression in Patients With De Quervain's Tenosynovitis; An Integrated Web Based Skills Intervention
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Data difficult to collect due to the COVID-19 pandemic.
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Neal Chung-Jen Chen, Interim Chief of the Hand & Arm Center, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2018P002064
Record Dates: First submitted 2019-08-16; First posted 2019-08-28 (Actual); Last update posted 2022-05-05 (Actual); Status verified 2022-04

CONDITIONS: De Quervain Disease
MeSH Terms: conditions — De Quervain Disease | interventions — Decision Support Techniques

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Usual care, no depression (Other): Participants without symptoms of depression who have the opportunity to use a Decision Aid but otherwise receive Usual care
  Interventions: Other: Decision Aid
- Usual care, depression (Other): Participants with symptoms of depression who are randomized to receive Usual care (in addition to the Decision Aid)
  Interventions: Other: Decision Aid
- Toolkit, depression (Active Comparator): Participants with symptoms of depression who are randomized to receive the Toolkit intervention in addition to Usual care
  Interventions: Other: Decision Aid; Behavioral: Toolkit for de Quervain's

INTERVENTIONS:
Other: Decision Aid — A website that contains information about de Quervain's tenosynovitis and the options for treatment
Behavioral: Toolkit for de Quervain's — A website that offers 4 sessions of mind-body skills to help manage pain from de Quervain's tenosynovitis
  Arms: Toolkit, depression

SUMMARY:
This study evaluates a Decision Aid to help patients with de Quervain's tenosynovitis decide how to treat their condition.

For patients with symptoms of depression, half the participants will receive a psychological intervention (Toolkit) to improve depression and pain from de Quervain's tenosynovitis.

The investigators hypothesize that both the Decision Aid and the Toolkit will be feasible, and that the Toolkit will improve pain and function compared to usual care.

DETAILED DESCRIPTION:
The investigators are doing this research to see if they can improve the management of patients with de Quervain's tendinopathy. In the first part of this study, a Decision Aid (DA) has been developed to help participants make choices about their treatment.

Decision aids are designed to provide patients with balanced, complete, and understandable information about their options for management of their condition, as well as risks and benefits, in order to help them determine their preferences according to their values. Research has shown that patients felt more knowledgeable and better informed with a more active role in decision making after using DAs.

Additionally, research has shown that depression affects pain and disability experienced by patients with de Quervain's tenosynovitis. In the second part of our study, the investigators want to see whether a web based skills intervention (Toolkit) is more effective than usual medical care in improving pain and disability in patients with de Quervain's tenosynovitis and symptoms of depression.

The Toolkit is delivered online and can be accessed at home. Similar skills interventions in patients with musculoskeletal injury have been shown to improve pain and function.

ELIGIBILITY:
Inclusion Criteria:

* Adults (≥18 years) diagnosed with de Quervain's tenosynovitis
* English fluency and literacy
* Ability to give informed consent

Exclusion Criteria:

* Inability or unwillingness to participate in decision aid (DA) and/or Toolkit-depression
* Major medical comorbidity expected to worsen in the next 6 months
* Comorbid chronic pain condition
* Antidepressant medications changes in the past 6 months
* Severe and untreated mental health conditions or active substance dependence
* Secondary gains such as litigations or worker compensation procedures that may interfere with patients' motivation for treatment
* No online device available to use the DA and Toolkit-depression

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2018-12-10 (Actual); Primary Completion 2022-02-19 (Actual); Study Completion 2022-02-19 (Actual)

PRIMARY OUTCOMES:
QuickDASH score (Disabilities of the Arm Shoulder and Hand) | 6 months
  This questionnaire measures individual's ability to complete daily tasks and the severity of their symptoms. The scoring scale ranges from 0 (no disability) to 100 (most severe disability).
Numerical Pain Rating Scale | 6 months
  This scale measures the patient's pain intensity. The scale ranges from 0 (no pain) to 10 (worst possible pain).

SECONDARY OUTCOMES:
Patient Health Questionnaire 9 | 6 months
  This questionnaire is used for screening and measuring the severity of depression. The scale ranges from 0 to 27 overall. A score between the range of 5-9 indicates minimal symptoms of depression. A score between 10-14 suggests minimal depression or mild, major depression. A range of 15-19 indicates moderately severe, major depression, and a score of greater than 20 suggests severe, major depression.
Pain Catastrophizing Scale | 6 months
  This scale measures the individual's level of catastrophic thinking related to pain. They are asked about the thoughts and feelings they have when experiencing pain. The responses range from 0 (not at all) to 4 (all the time). The total score ranges from O-52. There are three subscale scores that assess rumination, magnification, and helplessness. The helplessness score ranges from 0 (not helpless) to 24 (severe helplessness). The rumination score ranges from 0 (don't think about the pain) to 16 (constantly think about how much it hurts). The magnification score ranges from 0 (does not feel like the pain is or will be more serious) to 12 (thinks the pain will get more serious).

CONTACTS AND LOCATIONS:
Overall Officials: Neal C Chen, MD, Principal Investigator — Hand and Arm Center Lead, Massachusetts General Hospital; Ana-Maria Vranceanu, PhD, Principal Investigator — IBHCRP, Massachusetts General Hospital
Locations (1):
- Hand and Arm Center, Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-01-17): https://cdn.clinicaltrials.gov/large-docs/41/NCT04069741/Prot_SAP_001.pdf